CLINICAL TRIAL: NCT02161848
Title: Magnetic Resonance Imaging Study of Patients With Chronic Progressive External Ophthalmoplegia
Brief Title: MRI Study - Chronic Progressive External Ophthalmoplegia
Acronym: CPEO
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gitte Hedermann Pedersen, Bsc., Rigshospitalet, Denmark
Other Study IDs: H-3-2012-163 (CPEO)
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Progressive External Ophthalmoplegia
MeSH Terms: conditions — Ophthalmoplegia, Chronic Progressive External | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients: Patients with verified singe large-scale mtDNA deletions and chronic progressive external ophthalmoplegia.
  Interventions: Other: Magnetic Resonance Imaging
- Controls: Healthy controls matched for age and gender.
  Interventions: Other: Magnetic Resonance Imaging
- Patient group as Controls: Patients with mitochondrial DNA 3243A>G mutations
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — MRI of eye muscles, lower bag muscles, thigh muscles and calf muscles.

SUMMARY:
The purpose of this study is to investigate the fraction of fat on a MRI scan of lower bag muscles, thighs and calves in patients with the mitochondrial disease chronic progressive external ophthalmoplegia (CPEO).

Additionally an investigation of the volume of the eye muscles will be done and compared to the patient's clinical presentation of ptosis and ophthalmoplegia.

DETAILED DESCRIPTION:
The lack of energy and fatigue seen in patients with mitochondrial diseases have been assumed to be caused by an energy defect because of a genetic defect in the mitochondrial DNA.

The investigators have analyzed a few MRI scans of muscles from patients with CPEO and have seen an extended amount of fat in their muscles, which seems to progress with age. The patient's symptoms might be caused by the extended amount of fat and thereby a less amount of active muscle instead of the "energy defect".

This will be investigated in a group of patients with CPEO and the results will be compared with results from a group of healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Danish patients with verified single large-scale mtDNA deletions and chronic progressive external ophthalmoplegia.

Exclusion Criteria:

* Patients who have metal implants in the body, for instance surgical clips, cochlear implant, pacemaker etc.
* Patients who are pregnant or breast-feeding.
* Patients who are claustrophobic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Danish patients with verified single large-scale mtDNA deletions and chronic progressive external ophthalmoplegia.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Fat fraction in the muscles of the lower bag, thighs and calves | 1 day
  The investigators will make a 3-point Dixon scan of the muscles of the lower bag, thighs and calves and measure the fraction of fat in these muscles once per patient or control.

SECONDARY OUTCOMES:
Isokinetic muscle dynamometry of ankle flexion | 1 day
  Isokinetic muscle dynamometry of ankle flexion. This is made on a Biodex 3 and done once per patient or control the same day as the MRI-scan is done. These results are correlated with the amount of non-fat-infiltrated muscle on the MRI scans.
Isokinetic muscle dynamometry of ankle extension | 1 day
  Isokinetic muscle dynamometry of ankle extension. This is made on a Biodex 3 and done once per patient or control the same day as the MRI-scan is done. These results are correlated with the amount of non-fat-infiltrated muscle on the MRI scans.
Isokinetic muscle dynamometry of knee flexion. | 1 day
  Isokinetic muscle dynamometry of knee flexion. This is made on a Biodex 3 and done once per patient or control the same day as the MRI-scan is done. These results are correlated with the amount of non-fat-infiltrated muscle on the MRI scans.
Isokinetic muscle dynamometry of knee extension | 1 day
  Isokinetic muscle dynamometry of knee extension. This is made on a Biodex 3 and done once per patient or control the same day as the MRI-scan is done. These results are correlated with the amount of non-fat-infiltrated muscle on the MRI scans.

OTHER OUTCOMES:
MRI T1 scan of eye muscles | 1 day
  Investigation of the volume of the eye muscles on a MRI scan and compare these with the patients clinical presentation of ptosis and ophthalmoplegia. The MRI scan is done once per patient or control and at the same day as the other MRI scans.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Research Unit, Copenhagen, Denmark